CLINICAL TRIAL: NCT01110057
Title: A Randomised, Double Blind Study to Evaluate the Safety and Efficacy of the p38 Kinase Inhibitor, GW856553, in Subjects With Neuropathic Pain From Lumbosacral Radiculopathy
Brief Title: Efficacy Study in Lumbosacral Radiculopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113049
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Pain, Neuropathic
Keywords: p38 kinase inhibitor; male and female; patients
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): GW856553
  Interventions: Drug: GS856553
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo to match GW856553
  Arms: Placebo
Drug: GS856553 — GW586553 7.5mg bid
  Arms: Active

SUMMARY:
This study will be a double-blind, placebo-controlled, parallel group study. After enrolment and initial assessments, subjects will receive 35 days of study medication. During this treatment period, they will be randomised to either oral GW856553 7.5mg BID or matching placebo in a 1:1 ratio. Sufficient numbers of subjects will be recruited to obtain 128 evaluable subjects.

DETAILED DESCRIPTION:
This is a double-blind, randomised, placebo-controlled, parallel group study. Subjects will undertake a screening period which may last up to approximately 3 weeks, followed by a baseline period of 1 week, a randomised treatment period of 5 weeks and a follow-up period of approximately 2 weeks.

This is a multi-centre, double-blind, randomised, placebo-controlled study in subjects who have at least moderate intensity of neuropathic pain resulting from lumbosacral radiculipathy. It will investigate the efficacy, safety and tolerability of GW856553.

Approximately 142 subjects will be randomised to ensure 128 evaluable subjects. Randomisation ratio will be 1:1 for placebo or GW856553 respectively. The dose of GW856553 will be 7.5 mg BID.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects aged 18 - 80 years inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of:

Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea Child-bearing potential and agrees to use one of the contraception methods listed in the protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 14 days after the last dose of study medication. Male subjects must agree to use the contraception methods listed in the protocol

* A diagnosis of neuropathic pain due to lumbosacral radiculopathy with the following characteristics:
* Pain perceived in one or both lower limbs at sites consistent with the area innervated by the L4, L5 or S1 nerve roots, with or without other sensory symptoms in the affected areas; (typically, the pain may be perceived in the buttock, thigh, calf, leg, foot or toes).
* History of the pain suggestive that the cause of lumbosacral radiculopathy is due to injury of the lumbosacral nerve root(s) by degenerative disease of the vertebrae in the lumbosacral spine or associated soft tissues including the intervertebral discs, or secondary to spinal injury and not due to infection/abscess, haematoma or malignancy.
* Duration of pain should be at least 12 weeks since onset.
* Intensity of pain should be stable for the 2 weeks prior to Screening, based on clinical history.
* As part of the neurological examination, the investigator must also conduct the procedures specified in the Standardised Evaluation of Pain [Neuropathic Pain] (StEP) instrument [Scholz, 2009]2, and to calculate the total score. In the clinical opinion of the investigator, the diagnosis of lumbosacral radiculopathy should be supported by at least one of the following features at Screening or documented in the medical notes in relation to the current symptoms:

Pain/sensory disturbance in dermatomal/myotomal distribution precipitated or exacerbated by straight leg raising (the straight leg raising test should be performed as specified in StEP; Neurological examination of lower limbs shows impaired muscle power, sensory function or deep tendon reflexes in the territory of the affected nerve roots; The total StEP score is greater than 4 (indicative of lumbosacral radiculopathy as the cause of the pain); Electromyographic (EMG) evidence of denervation in muscles innervated by the affected nerve roots; Quantitative sensory tests (QST) showing evidence of altered sensory thresholds in dermatomes innerved by the affected nerve roots;

* At Screening, if the investigator is satisfied with the diagnosis based on clinical review, or if results from such investigations related to the current symptoms are already documented in the medical notes, then it is not essential for the investigator to conduct computerised tomography (CT)/magnetic resonance imaging (MRI), EMG or QST.
* It is a requirement for all eligible subjects to have the nature of their spinal disease established by imaging (CT/MRI) and reviewed by a neuroradiologist / Investigator prior to starting study medication. This CT/MRI should be reviewed by the Investigator to ensure that it is consistent with the clinical diagnosis without any of the aetiologies in the exclusion criteria
* Subjects on medications for neuropathic pain (may only be included in the study if they have been on stable doses of such medications for at least 4 weeks prior to baseline period (Day -7) and continue with such stable doses during the study.
* Subjects' baseline average daily pain score for neuropathic pain due to LSR on the PI-NRS, calculated as the average of their daily PI-NRS scores over the baseline period (Day -7 to Day -1), is greater than or equal to 4 on the PI-NRS, after wash-out of prohibited medications. Male subjects must agree to use the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 14 days after the last dose of study medication.
* Subject has provided full written informed consent prior to the performance of any protocol-specified procedure, which includes compliance with the requirements and restrictions listed in the consent form.

Key Exclusion Criteria:

* Subjects who, in the opinion of the Investigator, are unable to reliably delineate or assess their own pain by anatomical location/distribution (e.g. can the subject reliably tell the difference between their back pain and their lower limb pain and rate their intensity separately ?).
* Subjects with lumbar canal stenosis in which the pain in the lower limbs occur solely on walking and not at rest.
* Subjects with causes for their neuropathic pain other than that specified in the inclusion criteria [e.g. post-herpetic neuralgia, painful diabetic neuropathy, mononeuritis multiplex, central post-stroke pain, failed back surgery in relation to the presenting episode of radiculopathy, spinal abscess/infection/haematoma/malignancy, phantom limb pain, peripheral neuropathy due to alcoholism, malignancy, HIV, syphilis, drug abuse, vitamin B12 deficiency, hypothyroidism, liver disease, toxic exposure], pain associated with a substantial somatic pain component [e.g.non-neuropathic / musculoskeletal pain in lower limbs or other parts of the body apart from the back] or more than one cause or potential cause for pain symptoms or any concurrent rheumatic disease such as but not limited to fibromyalgia, rheumatoid arthritis or significant osteoarthritis. Any question regarding the acceptability of aetiology of the neuropathic pain should be discussed with the GSK medical monitor.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody or positive history of HIV.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* History of any liver disease within the last 6 months [with the exception of known Gilbert's disease].
* History of excessive regular alcohol consumption within 6 months of the study.
* History or presence of significant cardiovascular, gastro-intestinal, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs which, in the opinion of the Investigator may interfere with the study procedures or compromise subject safety.
* History or presence of any clinically significant abnormality in vital signs / ECG / laboratory tests, or have any medical or psychiatric condition, which, in the opinion of the Investigator, may interfere with the study procedures or compromise subject safety.
* Subject has clinical evidence of recent major depression (by medical history) except those subjects already controlled by anti-depressants at screening.
* Subjects who, in the clinical judgement of the investigator, may be malingering or be motivated by secondary gain from participation in the study, will be excluded.
* Unable to stop and remain abstained from non-pharmacological treatments for their neuropathic pain during the study
* History of hypersensitivity to GW856553 or its components thereof or a history of drug or other
* Pregnant or lactating females
* Subjects with conditions requiring immunosuppressive therapy, or otherwise considered immunosuppressed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2010-01-07 (Actual); Primary Completion 2010-08-23 (Actual); Study Completion 2010-08-23 (Actual)

PRIMARY OUTCOMES:
Change in average daily neuropathic pain score from Baseline up to Week 5 (Week 4 of double blind treatment) of treatment | Baseline (Day -7 to Day -1) and up to 5 weeks
  The scores were analyzed based on the 11 point Pain Intensity Numerical Rating Scale (PI-NRS) with 0 score indicating no pain and score of 10 indicating maximum pain. The adjusted mean values are represented as least square mean (LS mean) values.

SECONDARY OUTCOMES:
Change in average daily pain intensity rating score (PI-NRS) from Baseline (Day -7 to Day -1) to 5 Weeks | Baseline (Day -7 to Day -1) and up to 5 weeks
  A minimum of 500,000 samples were run and the number of times the treatment difference estimated as greater than 0 was recorded. Non-informative prior distributions were applied for each of the weeks' treatment difference. For each weekly pain score calculation, a minimum of 4 days or more was required. If less than 4 average daily pain scores were recorded for any given week; then, that week's pain score was considered as missing and was excluded from the statistical analysis. Reduction in pain intensity was calculated from pain intensity score at indicated week minus the baseline pain intensity score. The scores were analyzed based on the 11 point Pain Intensity Numerical Rating Scale (PI-NRS) with 0 score indicating no pain and score of 10 indicating maximum pain. Arithmetic mean values have been presented; however, statistical analysis has been presented for least square (LS) means.
Change in pain quality on the Short-Form McGill Pain Questionnaire (SF-MPQ) from Baseline up to 5 weeks. | Baseline (Day -7 to Day -1) and up to 5 weeks
  Pain intensities were produced for each of the 15 questions on the SF-MPQ, split by treatment group, dimension and date of assessment. The total number of missing responses were recorded. The Short Form McGill Pain Questionnaire has 15 questions with the first 11 questions representing the sensory dimensions and questions 12 onwards representing the affective dimensions. The total score will be derived as the sum of all 15 questions with sub-group scores calculated for each of the 2 different dimensions. Change from Baseline is the value at indicated time point minus the Baseline value.
Number of participants with intensities of pain by SF-MPQ method over 5 weeks | From Baseline (Day -7 to Day -1) up to 5 weeks
  The Short Form McGill Pain Questionnaire (SF-MPQ) has 15 questions with the first 11 questions representing the sensory dimensions and questions 12 onwards representing the affective dimensions. The total score was derived as the sum of all 15 questions with sub-group scores calculated for each of the 2 different dimensions. Data for few participants was not available (considered as missing). Based on intensity types of pain, participants with mild, moderate, severe and missing were considered.
Change in Galer Neuropathic Pain Scale score from Baseline up to Week 5 | Baseline (Day -7 to Day -1) and up to 5 weeks
  For the Galer neuropathic pain scale, the total score was calculated excluding question 8 with the maximum total score being 100. Higher scores indicated Worsening of pain. Supplementary to this, a sub score for non-allodynic pain was calculated from summing 8 items of the Galer Neuropathic Pain Score. The two items excluded from the sub score were those questioning sensitivity and surface pain, questions 6 and 10. Change from Baseline is the value at indicated time point minus the Baseline value. Arithmetic means have been presented; however, statistical analysis has been based on adjusted (LS) means.
Percentage of participants with more than or equal to (>=) 30% and >=50% reduction in average daily pain score relative to baseline up to 5 weeks | Baseline (Day -7 to Day -1) and up to 5 weeks
  The scores were analyzed based on the 11 point Pain Intensity Numerical Rating Scale (PI-NRS) with 0 score indicating no pain and score of 10 indicating maximum pain. The number of participants showing 30 percent and 50 percent reduction in average daily pain scores were recorded at Baseline (7 days prior to Day 1) on every Week up to 5 weeks. Change from Baseline is the value at indicated time point minus the Baseline value.
Percentage of participants who improved, much improved or very much improved relative to Baseline on the Patient Global Impression of Change (PGIC) and Clinical Global Impression of Change (CGIC) over 5 weeks | Baseline (Day -7 to Day -1) and up to 5 weeks
  The PGIC and CGIC are numeric scale and was meant to measure neuropathic pain that was measured on Days 8, 21 and 35 of treatment and the follow-up visit. The scale ranges from 0 to 7 with Very Much Improved=1, Much Improved=2, Minimally Improved=3, No Change=4, Minimally Worse=5, Much Worse=6, Very Much Worse=7. Lower scores indicated improvement and higher scores indicated worsening. PGIC scale was rated by participants and CGIC by respective clinicians. Change from Baseline is the value at indicated time point minus the Baseline value. The PGIC analysis was performed for low back pain.
Change in the score of the Oswestry Disability Index (ODI) from Baseline (Day -7 to Day -1) up to 5 weeks | Baseline (Day -7 to Day -1) and up to 5 weeks
  The Oswestry Disability Index consists of ten questions, each with a possible six answers. Each question was ranked from zero to five, with zero being showing no symptoms and five being the most severe case. The total score was derived for analysis by summing the individual responses from the ten questions, and dividing through by the total number of possible answers to the number of questions answered multiplied by 100. Change from Baseline is the value at indicated time point minus the Baseline value. Values were available only for Week 4 visit (Day 28).
Average total daily dose of rescue medication over 5 weeks | Up to 5 weeks
  Mean dose of rescue medication used to relieve pain was monitored over 5 weeks.
Change in total Profile of Mood States (POMS) score and POMS domains scores from Baseline to Weeks 3 and 5 of treatment | Baseline, Week 3 (Day 21), and Week 5 (Day 35)
  Profile of Mood States (POMS) questionnaire was used to assess a participant's mood over the previous week. It consists of 65 items, each with a score of 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a bit), and 4 (extremely). The item scores were summarized as a total score and also into 6 mood domain scores at each time-point. A higher score indicated a more negative mood state except for vigour which is weighted negatively and so a lower score indicates a more negative mood. The sum of each item in a domain was added together to get the overall domain score. The Mood Disturbance Total Score was obtained by summing up all 6 domains with the Vigour-Activity domain weighted negatively. If more than 2 scores are missing then the domain score was set to missing and for more than 4 items, the total score was not calculated. Change from baseline is the value at indicated time point minus the Baseline value.
Change in Sleep Interference Scale (SIS) from Baseline over 5 weeks | Baseline (Day -7 to Day -1) and up to 5 weeks
  Sleep interference score analysis was performed over 5 weeks. Change from Baseline is the value at indicated time point minus the Baseline value. Baseline was considered as 7 days prior to Day 1.
Change from Baseline (Day -7 to Day -1) in SF-36 Health over period | Baseline (Day -7 to Day -1) and Week 4
  The score from each question on the SF-36 was calculated by adding together each of the sub-questions. The overall total score was calculated as the sum over each of the 11 questions; however, for this study only questions 3 to 8 was completed and so the total score was based only on these questions. The different domains of SF-36 component have been described in the category titles. Change from Baseline is the value at indicated time point minus the Baseline value. Observed case (OC) data for only Week 4 was available and has been presented. Adjusted means have been presented as LS means.
Change in time to complete timed walk (20 m) from Baseline up to 5 weeks | Baseline (Day -7 to Day -1) and Week 4
  Participants were asked to walk for 20 meters at a pace they feel comfortable. When they had finished walking, they were instructed to record the intensity of their neuropathic pain again. The distance they had walked and the time taken was recorded. The change in intensity of pain after walking from before walking was defined as the walking-associated pain. Change from Baseline is the value at indicated time point minus the Baseline value. Median time required has been presented; however, the statistical analysis is based on the adjusted mean (LS mean) values. Data for only Week 4 is available and has been presented.
Change in walking-associated pain during timed walk from Baseline up to 5 weeks | Baseline and Week 4
  Participants were asked to walk for 20 meters at a pace they feel comfortable. When they had finished walking, they were instructed to record the intensity of their neuropathic pain again. The change in intensity of pain after walking from before walking was defined as the walking-associated pain. Change from Baseline is the value at indicated time point minus the Baseline value. Median time required has been presented; however, the statistical analysis is based on the adjusted mean (LS mean) values. Data for only Week 4 is available and has been presented.
Number of participants with death, adverse events (AEs) and serious adverse events (SAEs) | Up to 5 weeks
  Adverse event (AE) is an unfavorable change in the health of a participant, including abnormal laboratory findings, that happens during a clinical study or within a certain time period after the study has ended. This change may or may not be caused by the intervention being studied. Serious adverse event (SAE) is an adverse event that results in death, is life-threatening, requires inpatient hospitalization or extends a current hospital stay, results in an ongoing or significant incapacity or interferes substantially with normal life functions, or causes a congenital anomaly or birth defect. Medical events that do not result in death, are not life-threatening, or do not require hospitalization may be considered serious adverse events if they put the participant in danger or require medical or surgical intervention to prevent one of the results listed above.
Number of participants with vital signs outside the range of Potential Clinical Importance (PCI) | Up to 5 weeks
  Vital signs analyzed included diastolic blood pressure (DBP) , systolic blood pressure (SBP) ,and heart rate (HR). DBP more than (>) 100 millimeters of mercury (mm Hg) and <45 mm Hg was considered as of potentially clinical importance (PCI). SBP of >160 mm Hg and <85 mm Hg and HR of >110 beats per minute (bpm) and <40 bpm were considered of PCI.
Number of participants with abnormal electrocardiogram (ECG) findings over period | Up to 5 weeks
  Abnormal ECG values were recorded and were classified as abnormal and clinically significant (CS) and abnormal and not clinically /clinically insignificant (CI). The participants were analyzed over 5 weeks.
Number of participants with abnormal clinical chemistry, hematology, and urinalysis parameters over period | From Baseline up to 5 weeks
  Participants were analyzed for abnormality in clinical chemistry , hematological and urinalysis parameters over 5 weeks. Values were recorded abnormal as high (H) or low (L).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Denmark (2):
  - GSK Investigational Site, Hoersholm
  - GSK Investigational Site, Odense C
- France (5):
  - GSK Investigational Site, Bois-Guillaume
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
- Germany (4):
  - GSK Investigational Site, Schönau, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Hamburg
- Norway (3):
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Trondheim
- Sweden (2):
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113049 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register